CLINICAL TRIAL: NCT02520492
Title: Non Invasive Measurements of Intracranial Pressure in Patients With Malignant Glioma
Acronym: GMaPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: Laboratoire de Biophysique Neurosensorielle - UMR INSERM 1107 (Pr Paul AVAN) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01568-39
Record Dates: First submitted 2015-02-24; First posted 2015-08-13 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Glioma
Keywords: intracranial pressure
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- noninvasive method of ICP measurements (Experimental): Patients will receive a noninvasive measurement of ICP variations during each of their follow up consultation. These measurements will last until 30 minutes for the first consultation (parameters to determine) and 10 minutes for the others. A postural test will be performed during the ICP measurements when the patient condition will make it possible to do.
  Measurements will be performed by a device with noninvasive acoustic probes placed in the ear, and in case of electrophysiological test, regular electrodes on the brow.
  Interventions: Device: noninvasive method of ICP measurements (Elios)

INTERVENTIONS:
Device: noninvasive method of ICP measurements (Elios)
  Other Names: Elios device from ECHODIA company

SUMMARY:
In patients at risk of increased intracranial pressure (ICP), ICP measurements require invasive transducers, usually with insertion of a catheter into the cranium, or through a spinal tap. These invasive modalities involve risks and pain and they can be done only in specialized care units, with a high associated cost.

A novel method for detecting changes in ICP has developed recently. The auditory hair cells emit sounds and electric signals in response to sound, which can be easily detected and measured non-invasively with the help of a microphone probe placed in the external ear canal or regular electrodes. Indeed, the cochlear aqueduct connects the cerebrospinal fluid (CSF) spaces to the inner ear in such a way that ICP and inner-ear fluid pressure equalize within seconds.

A symptom of intracranial pressure (ICP) was observed in glioma patient due to a combination of causes: the inflammatory reaction around the tumor, the mass effect of the tumor, secondary vascular changes, a change in the flow of CSF.

The evaluation of intracranial hypertension by increased ICP (invasive) is not used in the monitoring of intracranial tumors. It is then detected by using routine clinical signs, in combination with a standard imaging method (MRI), but still subjective.

The measurement of noninvasive ICP could allow earlier detection of relapse, and evaluate whether the increase in ICP precedes tumor clinical worsening and / or imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant glioma who underwent a biopsy or a partial surgery of this tumor and a radiotherapy and/or chemotherapy treatment.
* Valid tympanometry test at least for one ear
* Between 18 and 65 years of age
* Cochlear response useful at least for an ear which has validate the tympanometry test
* Written informed consent reviewed and signed by patient
* Affiliation to a social security scheme

Exclusion Criteria:

* Patients who underwent a complete resection of their malignant glioma
* Invalid tympanometry test for the both ears
* Collect of cochlear responses impossible for the ear or both ear which validate the tympanometry test
* Patient refusal after enlightened information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04-03 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Presence of an ICP variation or increase when physician has diagnosed a clinical or morphological aggravation of the tumor with standard diagnose methods (composite outcome measure) | from baseline to 1 year
  Presence of an ICP variation or increase when physician has diagnosed a clinical or morphological aggravation of the tumor with standard diagnose methods (composite outcome measure ) : clinical signs, MRI and response assessment in neuro-oncology criteria (RANO) .

SECONDARY OUTCOMES:
evolution of ICP before and after the progression of the relapse tumor according to imaging (RMI) | from baseline to 1 year
evolution of ICP before and after the progression of the relapse tumor according to clinical sign | from baseline to 1 year
Evaluate efficiency of the measurement device of ICP changes on repetitive measurement as evaluated by composite outcome measure : clinical signs, MRI and RANO criteria | from baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, MD, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France

REFERENCES:
- [Derived] Casile M, Thivat E, Giraudet F, Ginzac A, Molnar I, Biau J, Brehant J, Lourenco B, Avan P, Durando X. Non-invasive intracranial pressure monitoring for high-grade gliomas patients treated with radiotherapy: results of the GMaPIC trial. Front Oncol. 2024 Jun 11;14:1302977. doi: 10.3389/fonc.2024.1302977. eCollection 2024. PMID 38919520